CLINICAL TRIAL: NCT02605811
Title: Radiation Versus Temozolomide in Preventing Brain Metastases in Limited Stage Small Cell Lung Cancer
Brief Title: Temozolomide in Preventing Brain Metastases in Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Haihong Yang, MD, Pricipal investigator, Associate Chief Physician, Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GACA1501
Record Dates: First submitted 2015-11-12; First posted 2015-11-16 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Small Cell Lung Cancer; Metastatic Carcinoma
Keywords: limited small cell lung cancer; brain metastases; prophylactic cranial radiotherapy; temozolomide
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma; Brain Neoplasms | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- temozolomide (Experimental): temozolomide oral 150mg/m2 d1-5/28d for 12 cycles
  Interventions: Drug: temozolomide
- prophylaxis cranial radiotherapy (Active Comparator): prophylaxis cranial radiotherapy,25-30Gy/10Fra
  Interventions: Radiation: prophylaxis cranial radiotherapy

INTERVENTIONS:
Drug: temozolomide
  Other Names: Temozolomide Capsules
  Arms: temozolomide
Radiation: prophylaxis cranial radiotherapy — 2
  Other Names: PCI
  Arms: prophylaxis cranial radiotherapy

SUMMARY:
To investigate the response of temozolomide versus prophylactic cranial radiotherapy in preventing brain metastases in completed or partial remission limited small cell lung cancer patients.

DETAILED DESCRIPTION:
We'd like to investigate the 2-year incidence rate of brain metastases in completed or partial remission limited small cell lung cancer patients who received temozolomide only for 12 months or 25-30Gy prophylactic cranial radiotherapy in preventing brain metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological diagnosis of small-cll lung cancer histology
2. 18 years or older
3. Eastern Cooperative Oncology Group (ECOG) Performance Status no more than 2
4. Local stage SCLC without distant metastases
5. After 1st-line chemotherapy (EP or IP) at least 4 cycles
6. After radical radiotherapy for primary tumor and lymph node drainage area:including concurrent or sequence chemoradiotherapy
7. CR or PR assessment by RECIST(1.0) before randomized
8. Haemoglobin 10.0 g/dl, Absolute neutrophil count (ANC) 1.5^9/L, platelets 100 x 10^9/L
9. Total bilirubin 1.5 x upper limit of normal (ULN) alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x ULN in the absence of liver metastases, or < 5 x ULN in case of liver metastases
10. Creatinine clearance 60ml/min (calculated according to Cockcroft-gault formula)

Exclusion Criteria:

1. Mixed non-small cell lung cancer histology
2. Neck and supraclavicular lymph node metastasis
3. Be allergic to temozolomide or intolerable to radiotherapy
4. Any unstable systemic disease
5. Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Estimated)
Dates: Start 2015-09; Primary Completion 2019-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
2-year incidence of brain metastases | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Hailing Yang, MD, Principal Investigator — the first affiliated hospital of Guangzhou MC
Locations (1):
- The first affiliated hospital of Guangzhou MC, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided